CLINICAL TRIAL: NCT05845242
Title: Image Features of LSCI and Thermography for Determining the Risk Factor (0,1,2 and 3) of Developing Diabetic Foot Ulcer
Status: Not yet recruiting | Type: Observational
Sponsor: Ziekenhuisgroep Twente (Other)
Collaborators: University of Twente (Other)
Responsible Party: Principal Investigator, KilianKappert, Principal Investigator, Ziekenhuisgroep Twente
Other Study IDs: ZGT_MYFOOT_LSCI
Record Dates: First submitted 2023-04-06; First posted 2023-05-06 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Diabetic Foot
Keywords: diabetic foot; diabetes; LSCI; thermography
MeSH Terms: conditions — Diabetic Foot; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Risk 0: Very low ulcer risk: No LOPS (loss of peripheral sensation) and No PAD (peripheral arterial disease)
- Risk 1: Low ulcer risk: LOPS or PAD
- Risk 2: Moderate ulcer risk: LOPS + PAD, or LOPS + foot deformity or PAD + foot deformity
- Risk 3: High ulcer risk: LOPS or PAD, and one or more of the following:
  * history of a foot ulcer
  * a lower-extremity amputation (minor or major)
  * end-stage renal disease

SUMMARY:
Diabetic foot ulcers are one of the complications of diabetes mellitus. These wounds are often the result of diabetes-related neuropathy and/or an ischemic foot. Even with great care, recurrent ulcers are common. To mediate the damage and societal costs that come with DF there is a need for applications to detect ulcers before they come apparent. Two of these promising techniques are Laser Speckle Contrast imaging and thermography. This study is part of 4 specific clinical studies and is aimed at determining Laser Speckle Contrast imaging and thermography features, the provocations that are needed to optimize imaging and the correlation between these features and the IWGDF risk stratification category system for the diabetic foot.

DETAILED DESCRIPTION:
Diabetic foot ulcers are one of the complications of diabetes mellitus. These wounds are often the result of diabetes-related neuropathy and/or an ischemic foot. Diabetic feet (DF) are ideally treated by a multidisciplinary wound care team. Patients at high risk and especially patients that suffer from DF before will have to be checked regularly for new wounds.

Even with great care, recurrent ulcers are common. To mediate the damage and societal costs that come with DF there is a need for applications to detect ulcers before they come apparent. To improve care, an application to predict the healing status is desired.

To this purpose, a set of four (4) specific clinical studies has been conceived to tackle the overall challenging objectives to characterise the risk of ulcers in different patients and through different measurement conditions, including conditions of how a tele-home care service can be deployed. This is clinical study A.

This study investigates two techniques:

Laser speckle contrast imaging (LSCI) is a promising non-invasive technique to assess microcirculation. LSCI, exploits the random speckle pattern that is generated when tissue is illuminated by laser light and changes when blood cells move in the sampled tissue.

Thermography is used to measure temperature distribution on the foot. It is expected that soon-to-be affected regions will be warmer than other regions. Also, regions with impaired blood supply can be recognized.

Clinical study A aims at determining Laser Speckle Contrast imaging and thermography features, the provocations that are needed to optimize imaging, and the correlation between these features and the IWGDF risk stratification category system for the diabetic foot.

ELIGIBILITY:
Inclusion Criteria:

* The sample will include all the people who sign the informed consent.
* Patients above 18. Patients diagnosed with Diabetic feet.
* Patients with Risk Level 0, 1, 2 and 3 according to the International Working Group on the Diabetic Foot - IWGDF).

Exclusion Criteria:

* People who do not give their consent to participate in the study.
* Patients with active wounds on one or both feet.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with diabetic foot, receiving check-ups at the out-patient clinic at ZGT in Almelo, The Netherlands.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2023-08-01 (Estimated); Primary Completion 2027-10-01 (Estimated); Study Completion 2028-10-01 (Estimated)

PRIMARY OUTCOMES:
Perfusion units at various regions of interest using LSCI | During one outpatient visit (30 minutes)
  Maps of perfusion units will be gathered for different risk groups. The perfusion units will be used to create risk features together with thermography .
Temperature at various regions of interest using thermography | During one outpatient visit (30 minutes)
  Maps of perfusion units will be gathered for different risk groups. The Temperature will be used to create risk features together with perfusion units from LSCI .
The effect of provocations performed prior to measuring with LSCI | During one outpatient visit (30 minutes)
  For both LSCI and thermography the circulation in the leg will be provoked using the leg raise maneuver or a pressure cuff. The effect on both measurements with and without these provocations will be evaluated.
The effect of provocations performed prior to measuring with thermography | During one outpatient visit (30 minutes)
  For both LSCI and thermography the circulation in the leg will be provoked using the leg raise maneuver or a pressure cuff. The effect on both measurements with and without these provocations will be evaluated.
Correlation of the above features with the chance of developing ulcers (Risk 0, Risk 1, Risk 2 and Risk 3). | Year 4
  A first attempt will be made to find a correlation between perfusion and temperature and how these differ depending on the risk factor.

SECONDARY OUTCOMES:
Gathering data for AI (artificial intelligence) risk factor analysis in MYFOOT study | Year 4
  Data will be gathered for other work packages in the consortium that focus on creating a model for clinical decision making.
Assessing the practical needs for transferring measurements to a different environment (e.g., home) by interviewing the clinicians involved in the consortium. | Year 3
  Other work packages in the greater MYFOOT consortium focus on transferring technologies from the hospital to the patient's home. Based on the workflow created in this study and the expert opinion of the clinicians involved in the consortium it will be decided if and how LSCI and thermography can be measured at a patient's home.

CONTACTS AND LOCATIONS:
Overall Officials: Kilian Kappert, PhD, Principal Investigator — ZGT